CLINICAL TRIAL: NCT04301323
Title: A Two-year, Randomized, Single-centre, Double-masked, Comparative Study to Evaluate the Annual Rate of Myopia Progression of Children With Myopia Receiving Daily BHVI1, BHVI2 Eye Drops Either Alone or in Combination
Brief Title: Myopia Control With Novel Eye Drops
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hai Yen Eye Care (Industry)
Collaborators: Brien Holden Vision Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS/AS/18/12; VCRTC-2018-02 (Other: HYEC-BHVI)
Record Dates: First submitted 2020-03-04; First posted 2020-03-10 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2021-08

CONDITIONS: Myopia
Keywords: Atropine; Combination eye drops; Myopia control
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: In the intervention group, there will be a minimum of 105 participants enrolled with the participants randomised to 3 groups of 35 in each group to receive either BHVI1, BHVI2 , or BHVI3 per group.
  In the non-randomized, matched control group, there will be 105 other participants recruited with similar inclusion and exclusion criteria and similar procedures as outlined but without any eye drops.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In the interventions group, the participants and the investigators will be masked to the nature of the drop dispensed. Upon receiving the product, the product will be coded and masked by a person other than the clinicians involved in the study. Only coded and masked product will be dispensed to the participant.
  Unmasking should only occur in the case of an adverse event if knowledge of the trial treatment would alter the plan of care for the participant. If at all possible (if time permits) the Sponsor / The Independent Pharmacist should be consulted prior to unmasking. Thorough documentation must occur, and exposure to treatment knowledge should be limited only to those who must know.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BHVI1 (Experimental): BHVI1 eye drops
  Interventions: Drug: BHVI1 eye drops
- BHVI2 (Experimental): BHVI2 eye drops
  Interventions: Drug: BHVI2 eye drops
- BHVI3 (Experimental): Combination of BHVI1 and BHVI2 eye drops
  Interventions: Drug: BHVI3 eye drops
- Non-randomized control group (No Intervention): a separate control group including 105 children enrolled and followed with only single-vision spectacles.

INTERVENTIONS:
Drug: BHVI1 eye drops — Including 35 children enrolled to receive BHVI1 eye-drops once nightly
  Other Names: Novel BHVI1 eye drops
  Arms: BHVI1
Drug: BHVI2 eye drops — Including 35 children enrolled to receive BHVI2 eye-drops once nightly
  Other Names: Novel BHVI2 eye drops
  Arms: BHVI2
Drug: BHVI3 eye drops — Including 35 children enrolled to receive BHVI3, combination of BHVI1 and BHVI2, eye-drops once nightly
  Other Names: Novel BHVI3 eye drops
  Arms: BHVI3

SUMMARY:
Myopia currently affects 30% of the world and by 2050, almost 50% of the world will be myopic based on conservative estimates.1 In 2050, this will equate to almost 5 billion people with myopia, and those with high myopia will total almost 1 billion.1 Due to the growing public health concerns surrounding myopia, including treatments for visual complications associated with high myopia, the resultant lost productivity and increased cost to society, a solution to ameliorate this issue is imperative.

Current treatment strategies cannot prevent myopia, and their ability to slow myopia progression is variable, ranging from 10% to 59%.2 Based on the meta-analysis between the different interventions for myopia control, atropine eye-drops were proved the most effective strategy.3 Atropine has been used in myopia control treatment over the last 30 years in many countries with no serious adverse events reported.4-6 Moreover, atropine, a non-selective antimuscarinic agent, has been regularly applied in multiple other ocular conditions with respect to the official FDA approvals.7 8 Regarding the myopia management, recent studies show the significant effect of low dose atropine in controlling the progression of spherical equivalent with the least side-effects such as photophobia and blurry near vision.9 However, the lack of substantial data in reducing the axial growth rate of low dose atropine proposes a need of either using higher dose of atropine or in combination with other pharmaceutical agent having such the effect.

We therefore aim to determine in a two-year clinical trial, the efficacy of the eye drops used in our clinical trial for its role in slowing progression of myopia.

DETAILED DESCRIPTION:
6.1. NULL HYPOTHESES

There is no difference in the rate of progression of myopia as determined by change in spherical equivalent refractive error over time between PX using test eye drops compared to PX in the control arm.

There is no difference in the rate of progression of myopia as determined by change in axial length over time between PX using test eye drops compared to PX in the control arm.

6.2. DESCRIPTION Statistical analysis is planned to commence on completion of trial monitoring and the submission of the data analysis request form. Any interim analysis will be conducted as described in this section unless a documented request is received from the Sponsor and approved by the trial PI.

Data stored in relational databases will be imported into SPSS / STATA software for statistical purposes. Data will be investigated for quality using range checks and frequency distribution. Underlying distributions of variables will be tested. In general, variables measured on an interval scale with a sufficiently large sample size will be considered to follow a normal distribution. Outputs from the statistical analysis such as statistical tables will be copied over to Excel. All statistical results will be reported in Excel format.

6.3. NUMBER OF PARTICIPANTS Prior studies indicated that the annual progression of refractive error in Asian children using single-vision spectacles was -0.70 ± 0.45D. Thus approximately a minimum of 35 successfully enrolled subjects are required in each study group in order to demonstrate a statistically significant 50% difference in myopia progression (0.35 ± 0.45D) between test and control groups at the 5% level of significance with 80% power, using a 2-tailed distribution and assuming 20% dropouts. The detectable difference of 0.35±0.45 equates to an effect size of 0.78. G*power was used to compute the sample size.

6.4. SIGNIFICANCE A p-value less than or equal to 5% will be considered to be statistically significant.

6.5. INTERIM ANALYSIS The clinical trial will employ at least one interim analysis. Statistical adjustments to the level of significance for interim analysis will be based on an alpha spending function where the information fraction of the annual data at the time of the interim analysis will be multiplied by 5%. However, the interim analysis used to justify the need for study termination will set the statistical significance to 1%.

6.6. ANALYSIS Participants who have commenced the clinical trial treatment will be included in the analysis dataset. Reasons and frequency distribution of participants discontinued at baseline will be reported. The analysis of efficacy variables such as subjective ratings will employ only scheduled and evaluable visits. The analysis of safety variables such as adverse responses will include all visits, including all unscheduled visits. The trial PI can request an analysis of only those participants who have completed the trial. The default type of analysis will follow an Intent-to-Treat principle. The analysis plan for each primary and secondary endpoint is described here.

6.6.1. Primary Endpoint: Myopic progression using cycloplegic spherical equivalent Spherical equivalent will be recorded on an interval scale as obtained directly from the instrument. Progression of spherical equivalent defined as the change from baseline for each participant-eye will be computed and summarised as means ± standard deviations for each visit. Progression will be analysed using the intent to treat principle by linear mixed model. This model will account for the intra-subject correlation due to eye specific data and repeated visits by using subject random intercepts. The fixed effects will include treatment groups and visits. Subjects will be factored as random effects. The model will also include confounding demographic factors and baseline readings to obtain unbiased estimates. Estimated means and its confidence limits will be reported based on the model.

Progression of spherical equivalent will also be converted to a binary format using a progression value such as -0.5D. Binary outcome variables will be analysed using logistic regression. Robust estimator of variance will be used to account for within subject correlation due to eye specific data.

6.6.2. Secondary Endpoint: Myopic progression based on axial length change Axial length will be recorded on an interval scale as obtained directly from the respective instruments. Progression of axial length defined as the change from baseline for each participant-eye will be computed and summarised as means ± standard deviations for each visit. Progression in axial length will be analysed using the intent to treat principle by linear mixed model. This model will account for the intra-subject correlation due to eye specific data and repeated visits by using subject random intercepts. The fixed effects will include treatment groups and visits. Subjects will be factored as random effects. The model will also include confounding demographic factors and baseline readings to obtain unbiased estimates. Estimated means and its confidence limits will be reported based on the model.

6.6.3. Adverse Events Adverse events will be recorded on a binary scale of 0 and 1, where 1 denotes the incidence of a new event. Data will be summarised as incidence over participant-time and as a percentage of participant or participant-eyes. Incidence of the event over participant or participant-eyes will be compared between trial groups using logistic regression.

6.6.4. Other Variables Data will be summarised as means ± standard deviations for variables measured on an interval scale and median ± interquartile range for ordinal variables and percentages for those that are categorical. Other commonly used tests of significance at each visit may include paired t-tests and group t-test for parametric data and Wilcoxon signed-rank test and rank sum test for non-parametric data. Test of other variables may also include Analysis of Variance (ANOVA) and repeated measures ANOVA to test for between-participant and within-participant factors. Test of other categorical variables may include McNemar's, Fisher's Exact and Chi-Square tests for within- and between-participant factors

6.6.5. Statistical Adjustments Difference between trial groups will be ascertained at the baseline visit. If there are significant differences, the baseline value can be used as a covariate adjustment in the statistical model. Difference from baseline can also be computed and used for further statistical analysis. If the differences are statistically significant, but of low clinical significance, the analysis can be conducted without these adjustments. However, the clinical relevance of the baseline differences will be discussed with the trial PI.

Simultaneous multiple group comparisons in a post-hoc analysis will be corrected using Bonferroni correction. No adjustments will be made for testing multiple endpoints such as multiple subjective ratings.

6.6.6. Deviations from Statistical Plan The end of study analysis will be conducted as described in the protocol. Any changes to this plan will be documented in the data analysis request form and will need to be duly authorised by the study principal investigator. The data analysis request form will be retained along with other study documentation.

6.7. SUB GROUP ANALYSIS The planned sub group analysis will be used only to investigate further hypotheses and not to make any conclusive inferences.

6.8. CRITERIA FOR TERMINATION OF THE TRIAL FOR FINAL DATA ANALYSIS The trial will be terminated upon completion of the final visit by the last active participant or if any of the conditions of Section 6.4 (Participant Withdrawal) are met. An active participant is one who is enrolled in the clinical trial and has not been discontinued.

6.9. PROTOCOL DEVIATION PROCESS AND ACCOUNTABILITY OF DATA

The clinical trial team will bring deviations to the attention of the PI who, pending the significance of the deviation, will discuss with the Biostatistician, and with the Sponsor, as required.

When applicable, at the end of each protocol, protocol deviations will be reviewed (masked) to determine whether any data should be excluded from the final analysis. A list of protocol deviations and a recommendation of the PI as to how to use the data collected at the respective visit will be given to the Sponsor for approval prior to data analysis.

Individual datapoints that are missing will be excluded from analysis involving only those specific variables. A participant's complete visit data will not be excluded if some of the observations are missing. Data from unscheduled visits will be used only for adverse response analysis. Inclusion of outliers in the analysis will be based on the magnitude of change in test statistics with and without the outliers. Outliers will preferably be retained unless there is significant change in test results.

The Clinical Ophthalmologist, in conjunction with the PI (Research Ophthalmologist), may label the clinic visit as "non evaluable" on any deviations as deemed appropriate. This would then be used to exclude the clinical trial visit from the analysis. Any other variable-specific exclusion will be listed in the analysis request form and approved by the trial PI.

A list is generated of all protocol deviations reported, and this information and any subsequent analysis and comment, is included in the final "Clinical Investigation - End of Clinical trial Report".

QUALITY CONTROL AND QUALITY ASSURANCE 7.1. CRTC MONITORING A monitor will ensure all essential documents are in place prior to study commencement and that all participants have signed the participant informed consent form prior to any study procedures being performed. No other monitoring will be performed due to the scale of the project.

7.2. PROTOCOL AMENDMENTS Protocol amendments will be submitted to the Sponsor and HREC for review and approval prior to implementation, unless the change required is to eliminate an immediate hazard to participants, or involves only administrative and/or logistical aspects of the studies (e.g. change in contact numbers).

7.3. PROTOCOL DEVIATIONS The Investigator will not deviate from the protocol except if the deviation affects Participants' rights, safety and well-being. Any deviation from the protocol shall be recorded together with an explanation, including corrective and preventive actions and reported to the required bodies within the specified timeframe. The Sponsor is responsible for analysing and assessing the significance of the deviation and determining if data will be excluded.

7.4. MAINTENANCE AND CALIBRATION OF EQUIPMENT Equipment will be monitored regularly for maintenance and calibration as per relevant Institute / CRTC SOPs, company and product manuals.

ETHICAL CONSIDERATIONS The protocols require HREC approval prior to start and will be conducted as per the applicable regulatory requirements.

The Investigator is to ensure that the protocol, PI/ICF, Investigator Brochure, available safety information, information about payment and compensation to participants, advertising or any clinical trial-specific information provided to participants (including potential participants), the Investigator's CV and/or evidence of appropriate qualifications and any other documentation they may request are submitted, reviewed and approved by the HREC. Any subsequent amendments will be reviewed and approved by an HREC prior to implementation.

8.1. CONFIDENTIALITY Confidentiality will be maintained throughout the studies by all parties involved in accordance with guidelines under Section 95 of the Privacy Act 1998, and guidelines approved under Section 95a of the Privacy Act 1998 (December 2001). Data will be secured against unauthorised access.

Privacy and confidentiality of information about each participant will be preserved in the reports and any publication of the clinical trial data.

8.2. INFORMED CONSENT The informed consent process and documentation to be used for the trial will be reviewed and approved by the HREC prior to use.

The informed consent process provides the participant with ongoing explanations that will allow them to make educated decisions about whether to begin or continue participating in the trial. The Investigator will discuss the trial with the participant and the participant will have the opportunity to ask questions before, during and after the trial. The participant will be informed that at any time during their involvement in the trial, they have the opportunity to withdraw this consent.

The PI/ICF provides a summary of the trial, including its purpose, procedures and schedule, potential risks and benefits, and alternative treatments. It also explains the participant's rights once in the trial. The participant is given sufficient time to consider whether or not to participate and if they agree to voluntarily take part, they give their consent by signing the PI/ICF.

ELIGIBILITY:
Inclusion Criteria: Subjects enrolled in the trial must:

* be accompanied by a parent or guardian who is able to read and comprehend Vietnamese/English and give informed consent as demonstrated by signing a record of informed consent;
* at baseline, be within the age range of 6 to 13 years old inclusive;
* be diagnosed as myopic having spherical equivalent between -0.50 diopter and-6.00 diopter.
* willing to comply with the applying eye drops once nightly at bedtime and follow the clinical trial visit schedule as directed by the Investigator.
* be willing to comply with the wearing and clinical trial visit schedule as directed by the investigator;
* have ocular findings deemed to be normal
* vision correctable to at least 20/25 or better in each eye with spectacles.

Exclusion Criteria: Subjects enrolled in the trial must NOT have:

* Any pre-existing ocular irritation, allergic conjunctivitis, injury or condition, including infection or disease.
* Any systemic disease that adversely affects ocular health e.g. diabetes, Graves disease, and auto-immune diseases such as ankylosing spondylitis, multiple sclerosis, Sjögrens syndrome and systemic lupus erythematosus. Conditions such as systemic hypertension and arthritis do not automatically exclude prospective participants.
* Use of or a need for concurrent category S3 and above ocular medication at enrolment and/or during the clinical trial.
* Use of or a need for any systemic medication or topical medications which may alter normal ocular findings / are known to affect a participant's ocular health / physiology or contact lens performance either in an adverse or beneficial manner at enrolment and/or during the clinical trial.
* NB: Systemic antihistamines are allowed on an "as needed basis", provided they are not used prophylactically during the trial and at least 24 hours before the clinical trial product is used.
* History of eye trauma
* History of use of myopia control interventions such as Orthokeratology or eye surgery.
* Contraindications to the products used in the trial such as pulmonary disease, heart conditions and ADHD
* Known allergy or intolerance to ingredients to eye-drops used in the trial and other related derivatives.
* Currently enrolled in another clinical trial.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2019-10-26 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Spherical equivalent | at baseline visit, at one-year and two-year visits
  Annual change in spherical equivalent from baseline

SECONDARY OUTCOMES:
Axial length | at baseline visit, at one-year and two-year visits
  Annual change in axial length from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Padmaja Sankaridurg, Professor, Study Director — Brien Holden Vision Institute; School of Optometry and Vision Science - University of New South Wales
Locations (1):
- Department of Ophthalmology - An Sinh Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Data would be available 6 months after the study ends and the study group could finalise the data analysis.

REFERENCES:
- [Background] Holden BA, Fricke TR, Wilson DA, Jong M, Naidoo KS, Sankaridurg P, Wong TY, Naduvilath TJ, Resnikoff S. Global Prevalence of Myopia and High Myopia and Temporal Trends from 2000 through 2050. Ophthalmology. 2016 May;123(5):1036-42. doi: 10.1016/j.ophtha.2016.01.006. Epub 2016 Feb 11. PMID 26875007
- [Background] Sankaridurg PR, Holden BA. Practical applications to modify and control the development of ametropia. Eye (Lond). 2014 Feb;28(2):134-41. doi: 10.1038/eye.2013.255. Epub 2013 Dec 6. PMID 24310242
- [Background] Huang J, Wen D, Wang Q, McAlinden C, Flitcroft I, Chen H, Saw SM, Chen H, Bao F, Zhao Y, Hu L, Li X, Gao R, Lu W, Du Y, Jinag Z, Yu A, Lian H, Jiang Q, Yu Y, Qu J. Efficacy Comparison of 16 Interventions for Myopia Control in Children: A Network Meta-analysis. Ophthalmology. 2016 Apr;123(4):697-708. doi: 10.1016/j.ophtha.2015.11.010. Epub 2016 Jan 27. PMID 26826749
- [Background] Brodstein RS, Brodstein DE, Olson RJ, Hunt SC, Williams RR. The treatment of myopia with atropine and bifocals. A long-term prospective study. Ophthalmology. 1984 Nov;91(11):1373-9. doi: 10.1016/s0161-6420(84)34138-0. PMID 6514306
- [Background] Shih YF, Chen CH, Chou AC, Ho TC, Lin LL, Hung PT. Effects of different concentrations of atropine on controlling myopia in myopic children. J Ocul Pharmacol Ther. 1999 Feb;15(1):85-90. doi: 10.1089/jop.1999.15.85. PMID 10048351
- [Background] Clark TY, Clark RA. Atropine 0.01% Eyedrops Significantly Reduce the Progression of Childhood Myopia. J Ocul Pharmacol Ther. 2015 Nov;31(9):541-5. doi: 10.1089/jop.2015.0043. Epub 2015 Jul 28. PMID 26218150
- [Background] Chatzistefanou KI, Mills MD. The role of drug treatment in children with strabismus and amblyopia. Paediatr Drugs. 2000 Mar-Apr;2(2):91-100. doi: 10.2165/00148581-200002020-00002. PMID 10937461
- [Background] Chen AM, Cotter SA. The Amblyopia Treatment Studies: Implications for Clinical Practice. Adv Ophthalmol Optom. 2016 Aug;1(1):287-305. doi: 10.1016/j.yaoo.2016.03.007. No abstract available. PMID 28435934
- [Background] Chia A, Lu QS, Tan D. Five-Year Clinical Trial on Atropine for the Treatment of Myopia 2: Myopia Control with Atropine 0.01% Eyedrops. Ophthalmology. 2016 Feb;123(2):391-399. doi: 10.1016/j.ophtha.2015.07.004. Epub 2015 Aug 11. PMID 26271839
- [Background] Fan DS, Lam DS, Chan CK, Fan AH, Cheung EY, Rao SK. Topical atropine in retarding myopic progression and axial length growth in children with moderate to severe myopia: a pilot study. Jpn J Ophthalmol. 2007 Jan-Feb;51(1):27-33. doi: 10.1007/s10384-006-0380-7. Epub 2007 Feb 9. PMID 17295137
- [Background] Kennedy RH, Dyer JA, Kennedy MA, Parulkar S, Kurland LT, Herman DC, McIntire D, Jacobs D, Luepker RV. Reducing the progression of myopia with atropine: a long term cohort study of Olmsted County students. Binocul Vis Strabismus Q. 2000;15(3 Suppl):281-304. PMID 11486796
- [Background] Yen MY, Liu JH, Kao SC, Shiao CH. Comparison of the effect of atropine and cyclopentolate on myopia. Ann Ophthalmol. 1989 May;21(5):180-2, 187. PMID 2742290
- [Background] Cooper J, Eisenberg N, Schulman E, Wang FM. Maximum atropine dose without clinical signs or symptoms. Optom Vis Sci. 2013 Dec;90(12):1467-72. doi: 10.1097/OPX.0000000000000037. PMID 24076540
- See also: Brien Holden Vision Institute — http://bhvi.org
- See also: Hai Yen Eye Care — http://haiyeneyecare.com
- See also: An Sinh Hospital — http://ansinh.com.vn
- See also: School of Optometry and Vision Science - University of New South Wales, Vietnam — http://www.optometry.unsw.edu.au/